CLINICAL TRIAL: NCT00769821
Title: The Impact of Lymphedema on Local and Overall Functioning
Brief Title: The Impact of Lymphedema on Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000616135; USCF-H452-29674-03; NCT00501436 (obsolete NCT alias)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer; Cancer Survivor; Lymphedema; Perioperative/Postoperative Complications
Keywords: lymphedema; perioperative/postoperative complications; cancer survivor; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: bioimpedance spectroscopy
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Gathering information from breast cancer survivors about lymphedema; its symptoms and their impact on shoulder, arm, and hand functioning; and quality of life may help doctors learn more about the disease.

PURPOSE: This clinical trial is studying the impact of lymphedema on breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the relationship between degree of lymphedema, lymphedema-associated symptoms, and local upper extremity functioning.
* To determine the relationship between degree of lymphedema, lymphedema-associated symptoms, local upper extremity functioning, and overall health-related functioning.
* To determine the relationship between degree of lymphedema, lymphedema-associated symptoms, local upper extremity functioning, overall health-related functioning, and quality of life.

OUTLINE: Patients are stratified according to presence of lymphedema (yes vs no).

Patients complete self-reporting questionnaires to assess the degree of lymphedema using the Norman Questionnaire and Jane M. Armer's Lymphedema and Breast Cancer Questionnaire; lymphedema-associated symptoms using Symptoms in the Affected Breast/Mastectomy site questionnaire, Symptoms in the Shoulder, Arm, or Hand on the Affected Side questionnaire, and General Symptom Experience questionnaire; local upper extremity functioning using hand dominance questionnaire and the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire; quality of life (QOL) using the Multidimensional QOL Scale; and comorbidity using the Charleston Comorbidity Scale. Patients undergo a 3.5-hour testing to assess the degree of lymphedema by arm circumference and bioimpedance spectroscopy (BIS); local upper extremity functioning by strength testing, range of movement and neurodynamic testing using a goniometer, a skin examination, skin sensation and sensation at scar using the Semmes-Weinstein Monofilament test, and fine motor control/finger coordination using the Purdue Pegboard, Finger Tapper, and Vibration Threshold; and overall health-related functioning using a graded exercise test.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * No breast cancer on both sides
  * No recurrence of breast cancer (local or distant)
* Completed active treatment for breast cancer (i.e., surgery and/or radiotherapy and/or chemotherapy) for ≥ 6 months

  * No prior contralateral or bilateral mastectomy
* No pre-existing lymphedema prior to breast cancer diagnosis
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Weight < 300 pounds
* Mentally and physically able to participate
* No current infection or lymphangitis involving the affected arm
* No pre-existing neuromuscular conditions that would affect local upper extremity or overall health-related functioning
* No contraindications to bioimpedance spectroscopy (BIS) testing, including the application of electrode adhesive pads to the skin (i.e., unable to lie supine, allergy to electrode adhesive pads, have sunburn, or have open wound)
* No contraindications to exercise testing as outlined by the American Heart Association and the American College of Sports Medicine

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2007-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Degree of lymphedema as assessed by the Norman Questionnaire, Jane M. Armer's Lymphedema and Breast Cancer Questionnaire, arm circumference, and bioimpedance spectroscopy (BIS) | study visit approximately 5 hours
Lymphedema-associated symptoms by Symptoms in the Affected Breast/Mastectomy site questionnaire; Symptoms in the Shoulder, Arm, or Hand on the Affected Side questionnaire; and General Symptom Experience questionnaire | study visit approximately 5 hours
Local upper extremity function by tests & questionnaires (e.g., hand dominance; strength; range of motion & neurodynamics; fine motor control/finger coordination; skin exam; skin & scar sensation [Semmes-Weinstein Monofilament]) | study visit approximately 5 hours
Overall health-related functioning as assessed by Medical Outcomes Study-Short Form 36 (MOS-SF36), graded exercise test using a treadmill stress test, and cardio-respiratory fitness using peak VO2 | study visit approximately 5 hours
Quality of life (QOL) as assessed by Multidimensional QOL Scale | study visit approximately 5 hours
Comorbidity as assessed by Charleston Comorbidity Scale | study visit approximately 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marylin J. Dodd, RN, PhD, FAAN, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco School of Nursing, San Francisco, California, United States